CLINICAL TRIAL: NCT00968591
Title: An Open-label, Single-dose Study to Assess the Pharmacokinetics of Oral Everolimus (Afinitor®) in Subjects With Impaired Hepatic Function
Brief Title: Pharmacokinetics of Everolimus in Subjects With Hepatic Insufficiency
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CRAD001X2102; EudraCT 2009-012295-27
Record Dates: First submitted 2009-08-27; First posted 2009-08-31 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2016-04

CONDITIONS: Hepatic Insufficiency
Keywords: Hepatic insufficiency; liver disease; cirrhosis; pharmacokinetics
MeSH Terms: conditions — Hepatic Insufficiency; Liver Diseases; Fibrosis | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RAD001 (Experimental)
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus

SUMMARY:
This clinical pharmacology research study will assess the safety and pharmacokinetics of the drug everolimus in patients with impaired hepatic function as compared to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

All subjects:

* In good health as determined by past medical history, physical examination, vital signs, electrocardiogram, and laboratory test values (except for values related to hepatic insufficiency).

Hepatic impaired subjects:

* A Child-Pugh Classification score clinically determined as Class A, Class B, or Class C.
* Absolute neutrophil count (ANC) > 1000 cells/mm3
* Hemoglobin > 9 mg/mL
* Platelet count > 50,000/mm3 at screening and baseline
* Serum creatinine ≤ 2.0 x ULN
* Free of significant medical disorders unrelated to the subject's hepatic disorder

Exclusion Criteria:

All subjects:

* Significant illness, including infections, or hospitalization within 4 weeks prior to dosing (hospitalization is allowed for hepatic impaired subjects if related to liver disease). Invasive systemic fungal infections need to be fully resolved prior to study entry.
* History of acute or chronic bronchospastic disease (including asthma and chronic obstructive pulmonary disease, treated or not treated).
* History of clinically significant drug allergy; history of atopic allergy (asthma, urticaria, eczematous dermatitis). A known hypersensitivity to the study drug (everolimus) or drugs similar to the study drug (other mTOR inhibitors, e.g., rapamycin or temsirolimus).
* Active bleeding during the last 28 days prior to dosing, including variceal bleeding.
* Except for hepatic impairment, any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs or which may jeopardize the subject in case of participation in the study.
* Use of tobacco within 7 days prior to dosing or during the study.
* Consumption of alcohol within 3 days prior to dosing or during the study.
* Consumption of grapefruits, grapefruit juice, Sevilla oranges, starfruit or related foods within 7 days prior to dosing or during the study period.
* Use of any drugs known to affect CYP3A4 or PgP, including both inhibitors and inducers, within 7 days prior to dosing or during the study.

Hepatic impaired subjects:

* Symptoms or history of Grade 3 or 4 hepatic encephalopathy within 4 weeks of study entry.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-11; Primary Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Evaluate the pharmacokinetics of a single oral dose of everolimus in subjects with severely impaired hepatic function (Child-Pugh C) relative to healthy controls. Measure: AUC, Cmax, tmax, λz, Vd/F, CL/F and t1/2 | First 8 days

SECONDARY OUTCOMES:
Evaluate the pharmacokinetics of a single oral dose of everolimus in subjects with mild and moderate impaired hepatic function (Child-Pugh A and B, respectively) relative to healthy controls. | First 8 days
Assess the safety and tolerability of a single oral dose of everolimus in subjects with impaired hepatic function (Child-Pugh A, B, and C). | First 8 days plus day 15 and day 28 post-dose follow-ups for safety
Explore correlation between pharmacokinetics and hepatic function parameters | First 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- Novartis Investigative Site, Frankfurt, Germany
- Novartis Investigative Site, Moscow, Russia
- Novartis Investigative Site, Singapore, Singapore

REFERENCES:
- [Derived] Peveling-Oberhag J, Zeuzem S, Yong WP, Kunz T, Paquet T, Bouillaud E, Urva S, Anak O, Sellami D, Kobalava Z. Effects of hepatic impairment on the pharmacokinetics of everolimus: a single-dose, open-label, parallel-group study. Clin Ther. 2013 Mar;35(3):215-25. doi: 10.1016/j.clinthera.2013.02.007. Epub 2013 Mar 1. PMID 23453404
- See also: Results for CRAD001X2102 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=4242